CLINICAL TRIAL: NCT00512291
Title: Study of Subcutaneous Olanzapine for Hyperactive or Mixed Delirium
Brief Title: Subcutaneous Olanzapine for Hyperactive or Mixed Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0746
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Hyperactive Delirium; Mixed Delirium; Olanzapine
MeSH Terms: interventions — Olanzapine; Fluoxetine; olanzapine-fluoxetine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olanzapine (Experimental): 5 mg subcutaneous injection every 8 hours for 9 doses
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — 5 mg subcutaneous injection every 8 hours for 9 doses. Each injection should take about 1 to 2 minutes.
  Other Names: Fluoxetine; Symbyax

SUMMARY:
The objective of this study is to determine the tolerability and safety of olanzapine administered as a subcutaneous injection to hospitalized patients with hyperactive or mixed delirium.

DETAILED DESCRIPTION:
Olanzapine is a drug designed to control agitation/delirium. Olanzapine has been given by mouth and as an injection into the muscle, which is painful and can increase a person's feelings of agitation. In this study, olanzapine will be given under the skin through a catheter. Researchers hope that this will be less painful and agitating than when injected into the muscle.

If you are found to be eligible to take part in this study, you will have a catheter (plastic tube) placed under your skin. This catheter will be used to give you the study medication. Study drug will be given through the catheter every 8 hours for 9 doses. Each shot should take about 1 to 2 minutes. You will receive the drug at M.D.Anderson Cancer Center.

Researchers will use the Richmond Agitation Scale to measure your agitation or sedation before each injection of olanzapine through the catheter. It should take 5 to 10 minutes to answer the questions. You will be evaluated for catheter site reaction at the time of injection, at 30 minutes and 1 hour after the injection, and before all further injections of study drug. Your blood pressure will be evaluated before and 1 hour after the first two injections and then once a day while on study.

If your agitation is not controlled, you will receive haloperidol. On the second day of treatment, researchers will record the amount of haloperidol that you had to use in the previous 24 hours. If the amount of haloperidol that you used is greater than a certain amount, your dose of olanzapine will be increased. Even if your dose of olanzapine is increased, you may still be able to use haloperidol if needed.

On the third day of treatment, researchers will record the amount of haloperidol that you had to use in the previous 24 hours. If the amount of haloperidol that you used is greater than a certain amount, your dose of olanzapine will again be increased. As before, if your dose of olanzapine is increased, you may still be able to use haloperidol if needed. If you respond to olanzapine after 3 days of treatment, you will be given the option to continue the drug off-study.

If you develop severe side effects before you have completed the 9 doses, treatment will be stopped. If treatment on this study is stopped, then you will consult with your doctor about receiving a different medication off study to help control your symptoms. There is no long-term follow-up for this study.

This is an investigational study. Olanzapine has been FDA approved given into the muscle or by mouth for the treatment of agitation related to schizophrenia and bipolar mania (a disorder involving mood swings from deep depression to feelings of elation). A total of 25 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients on the Acute Palliative Care Unit (G12NW) at the University of Texas MD Anderson Cancer Center
2. Age > 18 years of age (Olanzapine IM has not been evaluated in pediatric patients.)
3. Patients must have an acceptable surrogate capable of giving consent on the subject's behalf.
4. Richmond Agitation-Sedation Score (RASS) of >/= 1
5. Mini Mental Status Exam score of less than 24
6. Hyperactive or mixed delirium not responsive to at least 10 mg of haloperidol within the last 24 hours

Exclusion Criteria:

1. Known hypersensitivity to any ingredient of olanzapine IM
2. The following reactions to haloperidol: A) Acute dystonia B) Hypersensitivity or previous intolerance to haloperidol C) Extra pyramidal side effects
3. History of narrow-angle glaucoma.
4. Systolic blood pressure < 90 mm Hg
5. If they received an injectable depot neuroleptic within less than one dosing interval of study initiation
6. Within 7 days of starting study drug, documentation of: a. Fasting blood glucose (or finger stick glucose check) > 250 mg/dl b. Absolute neutrophil count of < 500 or platelets < 50,000
7. The use of any benzodiazepines or neuroleptic medications, besides haloperidol, while the patient is enrolled on study, is prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-06; Primary Completion 2007-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Participant Toxicity | Within 75 hours of the initial treatment
  Toxicity defined as urticaria, injection site reactions, and/or hypotension. At time 0, 0.5, and 1 hour after the first injection of study drug and prior to all subsequent injections of study drug, urticaria and injection site reaction assessed using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 3.0. Blood pressure evaluated immediately before and 1 hour after each of the first 2 injections, and then daily thereafter.
Participant Hypotension | 3 Days
  Participants who experience a drop in blood pressure below 90/50 mm Hg within 60 minutes post study drug administration. Blood pressure evaluated immediately before and 1 hour after each of the first 2 injections, and then daily thereafter.

SECONDARY OUTCOMES:
Participant Richmond Agitation Sedation Scale (RASS) | 3 Days
  Evaluation of RASS at time 0, once the injection is completed, at 0.5 hours post-injection, and at 1 hour post-injection for the first injection of study drug, and then prior to each injection of study drug to determine efficacy. Treatment efficacy defined as: RASS Score of less than 1 prior to the last dose on the third day; and Total haloperidol usage of less than 8 mg per day. Haloperidol amounts recorded for previous 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elsayem, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center official website — http://mdanderson.org